CLINICAL TRIAL: NCT00674843
Title: Phase 1 Study to Determine the Efficacy of Using Far Infrared Radiation to Manage or Treat Muscular Dystrophies.
Brief Title: The Efficacy of Using Far Infrared Radiation to Manage Muscular Dystrophies
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GAAD Medical Research Institute Inc. (Other)
Responsible Party: Dr. Kwasi Donyina/Founder and President, GAAD Medical Research Institute Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GAAD-MD-CTP1
Record Dates: First submitted 2008-05-06; First posted 2008-05-08 (Estimated); Last update posted 2009-08-17 (Estimated); Status verified 2009-08

CONDITIONS: Muscular Dystrophies
Keywords: MYOTONIC DYSTROPHY; MYOPATHIES; Distal Myopathies; Muscular Dystrophy, Duchenne; Phosphorylase Deficiency (McArdle Disease)
MeSH Terms: conditions — Muscular Dystrophies; Myotonic Dystrophy; Muscular Diseases; Distal Myopathies; Muscular Dystrophy, Duchenne; Glycogen Storage Disease Type V

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Radiation: Far Infrared Radiation (5μm to 20μm wavelength)
  Interventions: Radiation: Far Infrared Radiation

INTERVENTIONS:
Radiation: Far Infrared Radiation — Radiation: Far Infrared Radiation (5μm to 20μm wavelength) Far Infrared radiation for 30 to 40 minutes per treatment session.

SUMMARY:
The muscular dystrophies (MD) are a group of more than 30 neuromuscular disorders that are characterized by progressive skeletal muscle weakness, defects in muscle proteins and the death of muscle cells and tissue. This study will investigate the use of far infrared radiation for managing muscular dystrophies.

DETAILED DESCRIPTION:
Observations from our research studies indicate that, far infrared rays provide energy to the body, improve the autonomic functions of the nervous system, restore the functions of the endocrine system, strengthen the immune system, improve blood circulation and increase the level of oxygen in the cells and promote the regeneration of muscle cells, nerves and brain cells.

It is hereby postulated that irradiation using far infrared, with wavelength between 5 to 20 microns, of the central nervous system, the endocrine system and the whole body could prevent, control, manage or possibly cure these neuromuscular disorders.

ELIGIBILITY:
Inclusion Criteria:

* Persons with muscular dystrophies

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2008-05; Primary Completion 2010-05 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Management and Cure of muscular dystrophies | 2 Years

SECONDARY OUTCOMES:
Rehabilitation of people with muscular dystrophies | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Ken Nedd, M.D., Principal Investigator — GAAD Medical Research Institute Inc.
Locations (1):
- The Centre for Incurable Diseases, Toronto, Ontario, Canada